CLINICAL TRIAL: NCT00472251
Title: One-year Prospective Observational Study of BMI Change Effect of 5-alpha Reductase Inhibitor in Korean BPH Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry); Seoul National University Bundang Hospital (Other)
Responsible Party: Sang Eun Lee/Professor, Seoul National University Bundang Hospital
Other Study IDs: CRT110446
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: dutasteride; body mass index; testosterone
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is widely-accepted that serum testosterone level and BMI (body mass index) representative of the degree of obesity has negative correlation. Considering the fact that obesity is being mentioned as a risk factor for development of prostate cancer as well as other various life-threatening diseases (example: cardiovascular problems), the effect of BPH treatment agents on BMI is a subject that should certainly be elucidated. Meanwhile, to our knowledge, no prospective study has so far been performed on such issue in Asian population. Prior to generating hypothesis of the effect of 5 alpha reductase inhibitor on BMI, the real effect of 5 alpha reductase inhibitor on BMI change in Korean BPH patients has to be observed in real clinical practice. This study will test the effects of one-year medication of 5 alpha reductase inhibitor on BMI among Korean men with BPH.

DETAILED DESCRIPTION:
This study is a prospective, 1-year follow-up, observational study. We are planning to enroll 100 Korean patients with BPH. At each visit, patients' height, weight, abdominal circumference will be checked. Laboratory parameters including fasting glucose, HbA1c, serum testosterone, free testosterone, sex hormone-binding globulin, estradiol, maximum flow rate (measured by flowmetry) will be tested. Blood test will be performed twice (at baseline and at the end of study). 5mL of blood will be needed at each time from one subject. And total IPSS score will be evaluated after 1 year of treatment of 5 ARI. At every visit, use of above prohibited medicines and other medications will be investigated. In addition, any surgical procedures undertaken during study period will be asked and recorded.

Subjects of study will be allocated into 3 separate groups. Group 1 will be those taking 5 alpha reductase inhibitor (dutasteride) only for 1 year. Group2 will be those who switch from alpha blocker to dutasteride and take dutasteride for 1 year. Group 3 will be composed of those taking both alpha blocker and dutasteride for 1 year.

composed of

ELIGIBILITY:
Inclusion Criteria:

* Male patients with symptomatic BPH
* Prostate volume of 30 cm3 or greater measured by transrectal ultrasound
* International Prostatic Symptom Score(IPSS) of 9 or greater
* Maximum urinary flow rate (Qmax) of 15ml/s or less
* No definite evidence of prostate cancer (on transrectal ultrasound, DRE, or etc.)
* Given Informed consent

Exclusion Criteria:

* Post-void residual more than 250 mL
* History of cancer (including prostate cancer) or previous prostatic surgery
* Acute urinary retention within 3 months of enrollment
* Chronic alcohol abuser and heavy smoker (> 10 cigarettes/day)
* History of/current drug abuse including laxatives
* Any previous 5 ARI administration
* Type 1 DM or Type 2 DM regardless of treatment
* Clinically significant endocrine diseases at investigator's discretion including thyroid diseases.
* History of /current bulimia or anorexia nervosa
* Regular use of following prohibited medicines within 3 months prior to screening; A. Medicines which can affect salt/water retention such as diuretics, calcium channel blockers, gabapentin, pregabalin, etc B. Medicines which can affect body weight such as sibutramine, orlistat, phentermine, amphetamine, etc.

C. Anti-thyroid medication, thyroxine, cyproheptadine, tranquilizers, systemic corticosteroids, testosterone supplement, or other medications that are known to affect body weight or BMI

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited men aged 45-75 years with moderate to severe symptomatic BPH (IPSS > 7 and a peak urinary flow rate of < 15 mL/s),an enlarged prostate (≥30 mL on TRUS), a PSA level of <10 ng/mL, and no evidence of prostate cancer (on a DRE or TRUS) among patients who visited our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
body mass index | after 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Roehrborn CG, Lee M, Meehan A, Waldstreicher J; PLESS Study Group. Effects of finasteride on serum testosterone and body mass index in men with benign prostatic hyperplasia. Urology. 2003 Nov;62(5):894-9. doi: 10.1016/s0090-4295(03)00661-7. PMID 14624915